CLINICAL TRIAL: NCT00518713
Title: Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Clobazam in Patients With Lennox-Gastaut Syndrome
Brief Title: Clobazam in Patients With Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13110A; OV1012 (Other: Former study ID)
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-01

CONDITIONS: Epilepsy; Epilepsy, Generalized; Seizures
Keywords: Epilepsy; Lennox-Gastaut Syndrome; Drop seizures; Clobazam
MeSH Terms: conditions — Epilepsy; Epilepsy, Generalized; Seizures; Lennox Gastaut Syndrome; Syncope | interventions — Clobazam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clobazam Low Dose (Experimental)
  Interventions: Drug: Clobazam Low Dose
- Clobazam Medium Dose (Experimental)
  Interventions: Drug: Clobazam Medium Dose
- Clobazam High Dose (Experimental)
  Interventions: Drug: Clobazam High Dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clobazam Low Dose — 0.25 mg/kg/day; tablets; orally; for 15-18 weeks
  Other Names: Onfi™
  Arms: Clobazam Low Dose
Drug: Clobazam Medium Dose — 0.5 mg/kg/day; tablets; orally; for 15-18 weeks
  Other Names: Onfi™
  Arms: Clobazam Medium Dose
Drug: Clobazam High Dose — 1.0 mg/kg/day; tablets; orally; for 15-18 weeks
  Other Names: Onfi™
  Arms: Clobazam High Dose
Drug: Placebo — tablets; orally; daily for 15-18 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of clobazam as adjunctive therapy in the treatment of seizures which lead to drop attacks (drop seizures) in patients 2 to 60 years of age with Lennox-Gastaut Syndrome (LGS). Patients will be enrolled at approximately 65 sites in the U.S. and ex-US for up to 23 weeks. Patients will be randomly assigned to either a low, medium or high dose, or placebo. The study will include a baseline period, a titration period and a maintenance period. After the maintenance period, patients will either continue into an open-label extension study or enter the taper period with a final visit 1 week after the last dose.

DETAILED DESCRIPTION:
LGS poses a significant treatment challenge. No single antiepileptic drug (AED) provides satisfactory relief for all or most patients with LGS and a combination of treatments is often required. Even with combination therapy, many LGS patients show resistance to treatment. Adjunctive therapy with newer anticonvulsant medications has demonstrated efficacy for some patients, although polytherapy and high medication doses are often associated with unfavorable adverse event profiles.

More effective and better-tolerated treatment options are needed for this population of medically intractable epilepsy patients. Clobazam may provide an improved safety profile compared to other AEDs currently approved for the treatment of LGS and may have less hypotonia and drooling effects than other benzodiazepines.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been <11 years of age at the onset of LGS.
* Patient must have LGS.
* Patient must be on at least 1 AED.
* Parent or caregiver must be able to keep an accurate seizure diary.

Exclusion Criteria:

* Etiology of patient's seizures is a progressive neurologic disease. Patients with tuberous sclerosis will not be excluded from study participation, unless there is a progressive tumor.
* Patient has had an episode of status epilepticus within 12 weeks of baseline.
* Patient has had an anoxic episode requiring resuscitation within 6 months of screening.
* Patient has a clinically significant history of an allergic reaction or significant sensitivity to benzodiazepines.
* Patient is taking more than 3 concurrent AEDs.
* Patient has been on the ketogenic diet for less than 30 days prior to screening or suffers from frequent stooling.
* If the patient has a Vagal Nerve Stimulator (VNS), the settings have not been stable for at least 30 days prior to screening.
* Patient has taken corticotropins in the 6 months prior to screening.
* Patient is currently taking long-term systemic steroids (excluding inhaled mediation for asthma treatment) or any other daily medication known to exacerbate epilepsy. An exception will be made of prophylactic medication, for example, for idiopathic nephrotic syndrome or asthma.
* If the patient is taking felbamate, has been taking it for less than 1 year prior to screening.

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 238 (Actual)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (53):
- United States (34):
  - University of Alabama at Birmingham, Huntsville, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Childrens Hospital Los Angeles, Los Angeles, California
  - The Children's Hospital, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Pediatric Neurology and Epilepsy Center, Loxahatchee Groves, Florida
  - Child Neurology Center of NW FL, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Pediatric Epilepsy & Neurology Specialists, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Pediatric Neurology of Idaho Children's Specialty Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Kentucky, Kentucky Clinic, Department of Neurology, Lexington, Kentucky
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - The Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - Clinical Research Center of New Jersey (CRCNJ), Voorhees Township, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - University Neurology, Inc., Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Jefferson Epilepsy Center, Philadelphia, Pennsylvania
  - UTMG Pediatric Neurology, Memphis, Tennessee
  - Children's Medical Center at UT Southwestern-Dallas, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Baylor College of Medicine Pediatric Neurology, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (3):
  - Strategic Health Evaluators, Chatswood, New South Wales
  - Royal Melbourne Hospital Department of Neurology, Melbourne, Victoria
  - Austin & Repatriation Hospital (Austin Health) Epilepsy Research Centre, Melbourne, Victoria
- Vitebsk Regional Diagnostic Center, Vitebsk, Belarus
- India (14):
  - Neurology Center, Ahmedabad, Gujarat
  - St. John's Medical College Hospital, Bangalore, Karnataka
  - Malikatta Neuro Center, Mangalore, Karnataka
  - K. S. Hedge Medical Academy, Mangalore, Karnataka
  - Jaslok Hospital & Research Centre, Mumbai, Maharashtra
  - KEM Hospital & Research Centre, Pune, Maharashtra
  - P.D. Hinduja National Hospital Medical Research Centre, Mumbai, Mumbai
  - Maulana Azad Medical College and Associated Lok Nayak Govind Ballabh Pant Hospitals and Guru Nanak Eye centre, New Delhi, National Capital Territory of Delhi
  - Institute of Human Behaviour and Allied Sciences, Delhi, New Delhi
  - Deenanath Mangeshkar Hospital and Research Center, Erandawane, Pune
  - Christian Medical College, Ludhiana, Punjab
  - Dr. Kamakshi Memorial Hospital, Chennai, Tamil Nadu
  - Chhatrapati Sahu Ji Maharaj Medical University, Lucknow, Uttra Pradesh
  - Apollo Gleneagles Hospitals, Kolkata, West Bengal
- Kaunas University of Medicine Hospital, Kaunas, Lithuania

REFERENCES:
- [Result] Ng YT, Conry JA, Drummond R, Stolle J, Weinberg MA; OV-1012 Study Investigators. Randomized, phase III study results of clobazam in Lennox-Gastaut syndrome. Neurology. 2011 Oct 11;77(15):1473-81. doi: 10.1212/WNL.0b013e318232de76. Epub 2011 Sep 28. PMID 21956725
- [Derived] Brigo F, Jones K, Eltze C, Matricardi S. Anti-seizure medications for Lennox-Gastaut syndrome. Cochrane Database Syst Rev. 2021 Apr 7;4(4):CD003277. doi: 10.1002/14651858.CD003277.pub4. PMID 33825230
- [Derived] Gidal BE, Wechsler RT, Sankar R, Montouris GD, White HS, Cloyd JC, Kane MC, Peng G, Tworek DM, Shen V, Isojarvi J. Deconstructing tolerance with clobazam: Post hoc analyses from an open-label extension study. Neurology. 2016 Oct 25;87(17):1806-1812. doi: 10.1212/WNL.0000000000003253. Epub 2016 Sep 28. PMID 27683846

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Started | 58 | 62 | 59 | 59
Modified Intent-to-Treat Population | 53 | 58 | 49 | 57
Completed | 50 | 45 | 41 | 41
Not Completed | 8 | 17 | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo | Total
Number analyzed (Participants) | 58 | 62 | 59 | 59 | 238
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 48 | 49 | 48 | 193
  Between 18 and 65 years | 10 | 14 | 10 | 11 | 45
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.9 (7.24) | 14.1 (10.42) | 11.7 (8.48) | 13.0 (9.17) | 12.4 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 25 | 21 | 94
  Male | 36 | 36 | 34 | 38 | 144

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Number of Drop Seizures (12-week Maintenance Period).
Description: Number of drop seizures (average per week) was obtained from seizure diaries. The average drop in seizures per week for patients who did not complete the maintenance period was calculated based on the time from the beginning of the maintenance period to date of withdrawal.
Time Frame: 4-week baseline period and 12-week maintenance period
Population: Modified Intent-to-Treat (MITT) population
Measure: Least Squares Mean (Full Range); unit: Percent Reduction
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent Reduction | 41.2 [-119 to 100] | 49.4 [-262 to 100] | 68.3 [-39 to 100] | 12.1 [-374 to 100]
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Placebo; Analysis of covariance (ANCOVA) with the percent reduction in drop seizures as the dependent variable and treatment, pooled center, and baseline drop seizure rate as the independent variables. A step-down procedure used, starting with the high dose versus placebo; Test type: Superiority or Other; p = 0.0120, ANCOVA
Statistical Analysis 2: Comparison: Clobazam Medium Dose vs Placebo; ANCOVA with the percent reduction in drop seizures as the dependent variable and treatment, pooled center, and baseline drop seizure rate as the independent variables. A step-down procedure used, starting with the high dose versus placebo; Test type: Superiority or Other; p = 0.0015, ANCOVA
Statistical Analysis 3: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Percent Reduction in Number of Drop Seizures (First 4 Weeks of the 12-week Maintenance Period).
Description: as for outcome 1
Time Frame: 4-week baseline period and the first 4 weeks of the 12-week maintenance period
Population: MITT population
Measure: Least Squares Mean (Full Range); unit: Percent reduction
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent reduction | 47.8 [-103 to 100] | 58.9 [-147 to 100] | 71.0 [-58 to 100] | 18.6 [-106 to 100]
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0027, ANCOVA
Statistical Analysis 2: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA

3. Secondary Outcome: Percent Reduction in Number of Drop Seizures (Middle 4 Weeks of the 12-week Maintenance Period).
Description: as for outcome 1
Time Frame: 4-week baseline period and the middle 4 weeks of the 12-week maintenance period
Measure: Least Squares Mean (Full Range); unit: Percent reduction
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 52 | 53 | 44 | 47
Percent reduction | 44.1 [-36 to 100] | 38.8 [-433 to 100] | 64.9 [-125 to 100] | 21.1 [-284 to 100]
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1041, ANCOVA
Statistical Analysis 2: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2207, ANCOVA
Statistical Analysis 3: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0025, ANCOVA

4. Secondary Outcome: Percent Reduction in Number of Drop Seizures (Last 4 Weeks of the 12-week Maintenance Period).
Description: as for outcome 1
Time Frame: 4-week baseline period and the last 4 weeks of the 12-week maintenance period
Measure: Least Squares Mean (Full Range); unit: Percent reduction
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 51 | 46 | 42 | 44
Percent reduction | 31.8 [-477 to 100] | 56.0 [-228 to 100] | 68.0 [-117 to 100] | -0.1 [-948 to 100]
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1469, ANCOVA
Statistical Analysis 2: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0161, ANCOVA
Statistical Analysis 3: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0024, ANCOVA

5. Secondary Outcome: Percent of Patients Considered Treatment Responders Defined as Those With a >=25%, >=50%, >=75%, 100% Reduction in Drop Seizures (12-week Maintenance Period).
Description: as for outcome 1
Time Frame: 4-week baseline period and the 12-week maintenance period
Measure: Number; unit: Percent of responders
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent of responders
  ≥ 25% reduction | 34 [0.83 to 4.20] | 46 [1.61 to 9.59] | 41 [2.14 to 14.30] | 28
  ≥ 50% reduction | 23 | 34 | 38 | 18
  ≥ 75% reduction | 15 | 22 | 31 | 6
  100% reduction | 4 | 7 | 12 | 2
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Placebo; ≥ 25% reduction. ANCOVA with the percent reduction in drop seizures as the dependent variable and treatment, pooled center, and baseline drop seizure rate as the independent variables. A step-down procedure used, starting with the high dose versus placebo; Test type: Superiority or Other; p = 0.1324, ANCOVA
Statistical Analysis 2: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0026, ANCOVA
Statistical Analysis 3: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0004, ANCOVA
Statistical Analysis 4: Comparison: Clobazam Low Dose vs Placebo; ≥ 50% reduction. ANCOVA with the percent reduction in drop seizures as the dependent variable and treatment, pooled center, and baseline drop seizure rate as the independent variables. A step-down procedure used, starting with the high dose versus placebo; Test type: Superiority or Other; p = 0.3383, ANCOVA
Statistical Analysis 5: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p = 0.0159, ANCOVA
Statistical Analysis 6: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 7: Comparison: Clobazam Low Dose vs Placebo; ≥ 75% reduction. ANCOVA with the percent reduction in drop seizures as the dependent variable and treatment, pooled center, and baseline drop seizure rate as the independent variables. A step-down procedure used, starting with the high dose versus placebo; Test type: Superiority or Other; p = 0.0279, ANCOVA
Statistical Analysis 8: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.0010, ANCOVA
Statistical Analysis 9: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.0001, ANCOVA

6. Secondary Outcome: Percent of Patients Considered Treatment Responders Defined as Those With a >=25%, >=50%, >=75%, 100% Reduction in Drop Seizures (First 4 Weeks of the 12-week Maintenance Period).
Description: as for outcome 1
Time Frame: 4-week baseline period and the first 4 weeks of the 12-week maintenance period
Population: MITT
Measure: Number; unit: Percent of responders
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent of responders
  ≥ 25% reduction | 71.7 | 82.8 | 89.8 | 52.6
  ≥ 50% reduction | 47.2 | 72.4 | 77.6 | 31.6
  ≥ 75% reduction | 35.8 | 44.8 | 63.3 | 14.0
  100% reduction | 13.2 | 19.0 | 30.6 | 3.5

7. Secondary Outcome: Percent of Patients Considered Treatment Responders Defined as Those With a >=25%, >=50%, >=75%, 100% Reduction in Drop Seizures (Middle 4 Weeks of the 12-week Maintenance Period).
Description: as for outcome 1
Time Frame: 4-week baseline period and the middle 4 weeks of the 12-week maintenance period
Measure: Number; unit: Percent Responders
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent Responders
  ≥ 25% reduction | 64.2 | 65.5 | 75.5 | 50.9
  ≥ 50% reduction | 43.4 | 51.7 | 71.4 | 24.6
  ≥ 75% reduction | 28.3 | 34.5 | 59.2 | 12.3
  100% reduction | 9.4 | 15.5 | 26.5 | 5.3

8. Secondary Outcome: Percent of Patients Considered Treatment Responders Defined as Those With a >=25%, >=50%, >=75%, 100% Reduction in Drop Seizures (Last 4 Weeks of the 12-week Maintenance Period).
Description: as for outcome 1
Time Frame: 4-week baseline period and the last 4 weeks of the 12-week maintenance period
Measure: Number; unit: Percent Responders
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent Responders
  ≥ 25% reduction | 66.0 | 60.3 | 71.4 | 43.9
  ≥ 50% reduction | 45.3 | 50.0 | 67.3 | 29.8
  ≥ 75% reduction | 28.3 | 36.2 | 57.1 | 12.3
  100% reduction | 13.2 | 15.5 | 20.4 | 5.3

9. Secondary Outcome: Tolerance
Description: Study responders who have ≥50% reduction in their drop seizure rate during the first 4 or first 8 weeks of maintenance compared to the 4 week baseline period.
Time Frame: 4-week baseline period and first 4/first 8 weeks of the maintenance period
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Participants
  ≥ 50% reduction - first 4 weeks of maintenance | 25 | 42 | 38 | 18
  ≥ 50% reduction - first 8 weeks of maintenance | 23 | 38 | 38 | 20

10. Secondary Outcome: Investigator Global Evaluations of the Patient's Overall Change in Symptoms.
Description: The physician was asked to rate the patient's overall change in symptoms and overall change in seizure activity and Quality of Life since the beginning of clobazam treatment by checking "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", or "very much worse".
Time Frame: Week 15
Population: Those patients in the MITT population who completed a Physician Global Evaluation at Week 15.
Measure: Number; unit: participants
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 52 | 57 | 49 | 55
participants
  Very much improved | 4 | 10 | 8 | 3
  Much improved | 20 | 27 | 23 | 10
  Minimally improved | 13 | 9 | 8 | 13
  No change | 12 | 9 | 6 | 22
  Minimally worse | 2 | 2 | 3 | 6
  Much worse | 1 | 0 | 1 | 1
  Very much worse | 0 | 0 | 0 | 0

11. Secondary Outcome: Parent/Caregiver Global Evaluations of the Patient's Overall Change in Symptoms.
Description: The parent/caregiver was asked to rate the patient's overall change in symptoms and overall change in seizure activity and Quality of Life since the beginning of clobazam treatment by checking "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", or "very much worse".
Time Frame: Week 15
Population: Those patients in the MITT population who had a baseline and Week 15 parent/caregiver global evaluations were analyzed.
Measure: Number; unit: participants
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 57 | 49 | 55
participants
  Very much improved | 8 | 13 | 11 | 4
  Much improved | 14 | 19 | 18 | 10
  Minimally improved | 20 | 14 | 11 | 11
  No change | 8 | 7 | 4 | 21
  Minimally worse | 2 | 2 | 3 | 6
  Much worse | 0 | 2 | 2 | 3
  Very much worse | 1 | 0 | 0 | 0

12. Other Pre Specified Outcome: Percent Reduction in the Number of Non-drop Seizures.
Description: This outcome measure evaluated the percent reduction (average per week) in non-drop Seizures. Non-drop seizures were other seizures not meeting the drop seizure definition. Drop seizures were defined as a drop attack or spell (atonic, tonic or myoclonic) involving the entire body, trunk, or head that led to a fall, injury, slumping in chair, or head hitting surface or that could have led to a fall or injury, depending on the position of the patient at the time of the attack or spell.
Time Frame: 4-week baseline period and the 12-week maintenance period
Measure: Least Squares Mean (Full Range); unit: Percent reduction
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent reduction | -53.3 [-1627 to 100] | -3.3 [-1591 to 100] | 40.0 [-190 to 100] | -76.3 [-1477 to 97]
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7210, ANCOVA
Statistical Analysis 2: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2505, ANCOVA
Statistical Analysis 3: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0924, ANCOVA

13. Other Pre Specified Outcome: Percent Reduction of Total (Drop and Non-Drop) Seizures.
Description: This outcome measure evaluated the percent reduction in average weekly rate in total (drop and non-drop) seizures. Drop seizures were defined as a drop attack or spell (atonic, tonic or myoclonic) involving the entire body, trunk, or head that led to a fall, injury, slumping in chair, or head hitting surface or that could have led to a fall or injury, depending on the position of the patient at the time of the attack or spell. Non-drop seizures were other seizures not meeting the drop seizure definition.
Time Frame: 4-week baseline period and 12-week maintenance period
Measure: Least Squares Mean (Full Range); unit: Percent reduction
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Number analyzed (Participants) | 53 | 58 | 49 | 57
Percent reduction | 34.8 [-155 to 100] | 45.3 [-523 to 100] | 65.3 [-49 to 100] | 9.3 [-189 to 100]
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0414, ANCOVA
Statistical Analysis 2: Comparison: Clobazam Medium Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0044, ANCOVA
Statistical Analysis 3: Comparison: Clobazam High Dose vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: 19 weeks
Arm/Group | Clobazam Low Dose | Clobazam Medium Dose | Clobazam High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 3/58 | 6/62 | 5/59 | 2/59
Other Adverse Events (participants affected / at risk) | 42/58 | 55/62 | 45/59 | 40/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clobazam Low Dose (N=58) | Clobazam Medium Dose (N=62) | Clobazam High Dose (N=59) | Placebo (N=59)
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 2 | 1
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Myoclonic epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Depressed level of consciousness (Psychiatric disorders) | 0 | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Ultrasound abdomen abnormal (Investigations) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clobazam Low Dose (N=58) | Clobazam Medium Dose (N=62) | Clobazam High Dose (N=59) | Placebo (N=59)
Constipation (Gastrointestinal disorders) | 1 | 1 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 3 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3 | 4 | 3
Fatigue (General disorders) | 3 | 3 | 2 | 1
Irritability (General disorders) | 2 | 7 | 3 | 3
Pyrexia (General disorders) | 10 | 6 | 7 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 6 | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 8 | 8 | 6
Urinary tract infection (Infections and infestations) | 1 | 3 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 3
Blood bicarbonate decreased (Investigations) | 1 | 0 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 4 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3 | 0
Ataxia (Nervous system disorders) | 2 | 1 | 6 | 2
Drooling (Nervous system disorders) | 0 | 8 | 8 | 2
Dysarthria (Nervous system disorders) | 1 | 1 | 3 | 0
Lethargy (Nervous system disorders) | 6 | 3 | 9 | 3
Psychomotor hyperactivity (Nervous system disorders) | 2 | 2 | 3 | 2
Sedation (Nervous system disorders) | 1 | 2 | 5 | 2
Somnolence (Nervous system disorders) | 9 | 15 | 15 | 7
Tremor (Nervous system disorders) | 1 | 4 | 1 | 0
Aggression (Psychiatric disorders) | 2 | 5 | 8 | 3
Insomnia (Psychiatric disorders) | 1 | 3 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review and approve all proposed abstracts, manuscripts, or presentations regarding this study prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.